CLINICAL TRIAL: NCT00685750
Title: Analysis of the Expression of a Specific Set of Genes and Tumor Antigens in Patients With Non-small Cell Lung Cancer or Melanoma
Brief Title: Expression Analysis of Specific Markers in Non-small Cell Lung Cancer or Melanoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrolment over the last 2 years with none in the past 1 year. No increase in the number of completed subjects for 1 year and no more ongoing study subjects
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 109752
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: tumor antigen; biomarkers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

ARMS (7):
- ME1 (Other): Patients with cutaneous metastatic melanoma receiving dacarbazine or temozolomide as first line treatment
  Interventions: Procedure: Collection of tumor and blood samples
- ME2 (Other): Patients with cutaneous metastatic melanoma receiving first line treatment other than dacarbazine or temozolomide only
  Interventions: Procedure: Collection of tumor and blood samples
- ME3 (Other): Patients with cutaneous metastatic melanoma receiving any second-or higherline chemotherapy treatment
  Interventions: Procedure: Collection of tumor and blood samples
- ME4 (Other): Patients with cutaneous metastatic melanoma receiving local irradiation of cutaneous/subcutaneous tumor lesions
  Interventions: Procedure: Collection of tumor and blood samples
- ME5 (Other): Patients with cutaneous metastatic melanoma receiving local imiquimod
  Interventions: Procedure: Collection of tumor and blood samples
- NSC (Other): Non-small cell lung cancer patients
  Interventions: Procedure: Collection of tumor and blood samples
- ME6 (Other): Patients with cutaneous metastatic melanoma receiving ipilimumab
  Interventions: Procedure: Collection of tumor and blood samples

INTERVENTIONS:
Procedure: Collection of tumor and blood samples — Samples will be collected before and after standard treatment

SUMMARY:
This study intends to analyze the expression of specific sets of markers in tumor samples and in serum from patients with Non-Small Cell lung Cancer (NSCLC) or Stage III or IV melanoma. The data obtained in this study will be used to guide future development of immunotherapies for melanoma or NSCLC patients. Moreover, the analyses will contribute to definition of markers potentially predictive of clinical response to specific anticancer therapies.

DETAILED DESCRIPTION:
This protocol posting has been updated due to a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* The patient (male or female) is at least 18 years of age.
* The investigator believes that the patient can and will comply with the requirements of the protocol.
* The patient has given his/her written informed consent to take part in the study.
* The investigator believes that it will be possible to obtain a tumor tissue sample of at least 3 mm3 before treatment and all required tumor tissues several weeks after the initiation of the treatment.
* The patient has cancer in one of the following histological types, fulfilling all of the characteristics listed for the respective cancer type:

Cutaneous Melanoma, unresectable stage III or stage IV • The patient has histologically documented unresectable stage III or stage IV metastatic cutaneous melanoma.

AND

• The patient is a candidate for one of the following treatments:

* First-line chemotherapy with DTIC or TMZ as monotherapy [group ME1],
* First-line chemotherapy with an agent other than DTIC/TMZ as monotherapy or a combination (that may, but need not, include DTIC, TMZ, IL-2 or IFNγ) [group ME2],
* Second- or higherline chemotherapy with any agent or combination of agents (that may, but need not, include DTIC, TMZ, IL-2 or IFNγ ; i.e., systemic chemotherapy after isolated limb perfusion should be considered as second-line) [group ME3],
* Palliative irradiation of skin lesion(s)/region, irrespective of what line of treatment is planned [group ME4],
* Topical palliative treatment by imiquimod of skin lesion(s), irrespective of what line of treatment is planned [group ME5].
* First or higher line treatment with ipilimumab [group ME6].

NSCLC, any stage if the patient is eligible for neo-adjuvant chemotherapy with subsequent resection • The patient has NSCLC at any stage (as defined by the International Staging System) if the patient is eligible for neo-adjuvant chemotherapy with subsequent resection.

AND

• The patient is a candidate for chemo(radio)-therapy induction doublet neoadjuvant chemotherapy with platinum plus a second chemotherapy drug.

[Note: Induction radiotherapy is permitted.]

The recruitment of patients to the NSCLC group has been ended prematurely.

Exclusion Criteria:

* The patient has any family history of congenital or hereditary immunodeficiency.
* The patient has in the two weeks before baseline received any of the following:
* Chemotherapeutic agents,
* Immune-modulating agents such as (but not confined to) IFN-α, IL-2, BCG and anti-cancer therapeutic vaccines,
* Immunosuppressive agents such as corticosteroids [except for prednisone, or equivalent, <0.5 mg/kg/day (absolute maximum 40 mg/day, maximum duration of treatment three weeks), and inhaled and topical steroids, which are allowed].
* The patient is currently receiving an anti cancer treatment in another clinical trial. However, if the patient has finished the drug administration phase of that trial and has entered the follow-up phase, this patient can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-04-28 (Actual); Primary Completion 2013-12-17 (Actual); Study Completion 2013-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (4):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Murray, Utah
- France (6):
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (16):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Ostercappeln, Lower Saxony
  - GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Hemer, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (4):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Padua, Veneto
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm

RESULTS

PARTICIPANT FLOW:
Groups:
- Melanoma 1 Group: Patients with cutaneous metastatic melanoma receiving nothing other than standard of care treatment consisting of dacarbazine or temozolomide as first line treatment
- Melanoma 2 Group: Patients with cutaneous metastatic melanoma receiving nothing other than standard of care treatment consisting of first line treatment other than dacarbazine or temozolomide only
- Melanoma 3 Group: Patients with cutaneous metastatic melanoma receiving nothing other than standard of care treatment consisting of any second-or higherline chemotherapy treatment
- Melanoma 4 Group: Patients with cutaneous metastatic melanoma receiving nothing other than standard of care treatment consisting of local irradiation of cutaneous/subcutaneous tumor lesions
- Melanoma 5 Group: Patients with cutaneous metastatic melanoma receiving nothing other than standard of care treatment consisting of local imiquimod
- Melanoma 6 Group: Patients with cutaneous metastatic melanoma receiving nothing other than standard of care treatment consisting of ipilimumab
- Non-Small Cell Group: Non-small cell lung cancer patients nothing other than any standard of care treatment.
Period: Overall Study
Arm/Group | Melanoma 1 Group | Melanoma 2 Group | Melanoma 3 Group | Melanoma 4 Group | Melanoma 5 Group | Melanoma 6 Group | Non-Small Cell Group
Started | 17 | 3 | 21 | 2 | 15 | 20 | 10
Completed | 17 | 3 | 19 | 2 | 15 | 20 | 9
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Tumor sampling failure | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Patient didn't receive the treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melanoma 1 Group | Melanoma 2 Group | Melanoma 3 Group | Melanoma 4 Group | Melanoma 5 Group | Melanoma 6 Group | Non-Small Cell Group | Total
Number analyzed (Participants) | 17 | 3 | 21 | 2 | 15 | 20 | 10 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (12.1) | 50.7 (12.5) | 64.5 (11.5) | 77.0 (5.7) | 65.5 (13.5) | 61.8 (16.7) | 59.5 (9.7) | 63.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 9 | 0 | 9 | 11 | 2 | 45
  Male | 6 | 0 | 12 | 2 | 6 | 9 | 8 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Expression of Tumor Antigens
Description: The outcome presents the number of participants with expression of MAGE-A3 and NY-ESO-1 tumor antigens, after administration of standard of care treatment course compared to before administration
Time Frame: Before and after administration of standard of care treatment course, up to 3 months
Population: The analysis was performed on the Total Treated cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma 1 Group | Melanoma 2 Group | Melanoma 3 Group | Melanoma 4 Group | Melanoma 5 Group | Melanoma 6 Group | Non-Small Cell Group
Number analyzed (Participants) | 17 | 3 | 21 | 2 | 15 | 20 | 10
Participants
  MAGE-A3: Remained Positive | 8 | 0 | 11 | 1 | 5 | 6 | 1
  MAGE-A3: Remained negative | 7 | 0 | 0 | 0 | 5 | 6 | 5
  MAGE-A3: Turned Positive | 0 | 0 | 0 | 0 | 1 | 1 | 0
  MAGE-A3: Turned Negative | 0 | 2 | 9 | 0 | 2 | 3 | 2
  MAGE-A3: Not tested | 1 | 0 | 0 | 1 | 2 | 1 | 0
  MAGE-A3: Invalid testing | 1 | 1 | 1 | 0 | 0 | 3 | 2
  NY-ESO-01: Remained Positive | 4 | 1 | 2 | 1 | 4 | 4 | NA — NY-ESO-01 gene signature was not assessed in this group
  NY-ESO-01: Remained negative | 9 | 1 | 14 | 0 | 6 | 11 | NA — NY-ESO-01 gene signature was not assessed in this group
  NY-ESO-01: Turned Positive | 1 | 0 | 1 | 0 | 1 | 1 | NA — NY-ESO-01 gene signature was not assessed in this group
  NY-ESO-01: Turned Negative | 0 | 0 | 1 | 0 | 2 | 0 | NA — NY-ESO-01 gene signature was not assessed in this group
  NY-ESO-01: Not tested | 2 | 0 | 2 | 1 | 2 | 1 | NA — NY-ESO-01 gene signature was not assessed in this group
  NY-ESO-01: Invalid testing | 1 | 1 | 1 | 0 | 0 | 3 | NA — NY-ESO-01 gene signature was not assessed in this group

2. Primary Outcome: Number of Subjects With a Pre-identified Gene Signature (GS) to the recMAGE-A3 Cancer Immunotherapeutic
Description: The outcome presents the number of participants with a pre-identified gene signature (GS) to the recMAGE-A3 cancer immunotherapeutic from before and after standard cancer treatment, for comparison.
Time Frame: Before and after administration of standard of care treatment course, up to 3 months
Population: The analysis was performed on the Total Treated cohort. Data was not collected for the subjects in Non-Small Cell Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma 1 Group | Melanoma 2 Group | Melanoma 3 Group | Melanoma 4 Group | Melanoma 5 Group | Melanoma 6 Group
Number analyzed (Participants) | 17 | 3 | 21 | 2 | 15 | 20
Participants
  Remained positive | 4 | 0 | 4 | 0 | 4 | 6
  Remained Negative | 9 | 0 | 7 | 0 | 3 | 5
  Turned Positive | 0 | 1 | 2 | 0 | 4 | 2
  Turned Negative | 1 | 1 | 1 | 1 | 1 | 4
  Not tested | 2 | 0 | 6 | 1 | 3 | 0
  Invalid testing | 1 | 1 | 1 | 0 | 0 | 3

3. Primary Outcome: The Serum Proteome
Time Frame: After administration of standard of care treatment course
Population: Proteome analysis on serum samples was not performed, because they, as a consequence of the early study termination, would not have added any scientific value and would not have benefited any individual patient.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 0

4. Primary Outcome: Correlation of Relevant Markers of the Pre-identified Gene-expression Signature as Measured by Immunohistochemical Methods and by Quantitative PCR.
Time Frame: After administration of standard of care treatment course
Population: The testing was not be performed, because, as a consequence of the early study termination, no scientific value would have been brought and no patient would have benefited from it.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 0

5. Primary Outcome: Number of NSCLC Patients With Gene-expression Signature and Tumor Antigens in Distinct Concomitant Tumor Lesions Obtained at the Same Time From the Same Patient.
Time Frame: After administration of standard of care treatment course
Population: as for outcome 4
Arm/Group | Overall Study Group
Number analyzed (Participants) | 0

6. Primary Outcome: Number of Patients Responding to Treatment, by Best Clinical Response Type
Description: This outcome was assessed for metastatic melanoma patients treated with ipilimumab, in order to explore the predictive value to clinical activity of pre-identified immune-related gene-expression signature, by evaluating the patient's best clinical response to this treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); POD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions.
Time Frame: At 6 months after the initiation of the ipilimumab therapy
Population: The analysis was performed on all the 25 subjects in the ME6 group that were tested for GS expression at Visit 1.
Measure: Count of Participants; unit: Participants
Groups:
- GS-positive Group: Patients with cutaneous metastatic melanoma receiving ipilimumab and who tested positive for Gene Signature expression at Visit 1.
- GS-negative Group: Patients with cutaneous metastatic melanoma receiving ipilimumab and who tested negative for Gene Signature expression at Visit 1.
- GS-invalid Group: Patients with cutaneous metastatic melanoma receiving ipilimumab and who had invalid tests for Gene Signature expression at Visit 1.
Arm/Group | GS-positive Group | GS-negative Group | GS-invalid Group
Number analyzed (Participants) | 14 | 10 | 1
Participants
  Complete response | 0 | 0 | 0
  Partial response | 1 | 0 | 0
  Stable Disease | 3 | 4 | 1
  Progressive Disease | 9 | 4 | 0
  Not evaluable | 1 | 2 | 0

ADVERSE EVENTS:
Description: No products under investigation were used in this study. As a result, there was no collection of adverse events during this study. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Melanoma 1 Group | Melanoma 2 Group | Melanoma 3 Group | Melanoma 4 Group | Melanoma 5 Group | Melanoma 6 Group | Non-Small Cell Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely and, as a consequence, all the study objectives were not fully assessed as specified in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.